CLINICAL TRIAL: NCT03790358
Title: Mood Effects of Serotonin Agonists
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 15-1311
Record Dates: First submitted 2018-12-21; First posted 2018-12-31 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Healthy
MeSH Terms: interventions — Lysergic Acid Diethylamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Lysergic Acid Diethylamide
- low dose MDMA (Experimental): 6.5ug dose of serotonin agonist
  Interventions: Drug: Lysergic Acid Diethylamide
- medium dose (Experimental): 13ug dose of serotonin agonist
  Interventions: Drug: Lysergic Acid Diethylamide
- high dose (Experimental): 26ug dose of serotonin agonist
  Interventions: Drug: Lysergic Acid Diethylamide

INTERVENTIONS:
Drug: Lysergic Acid Diethylamide — Drug will be administered in solution form.

SUMMARY:
The purpose of this study is to determine the effects of very low doses of serotonergic agonists on depressed mood in human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* English fluency
* High school level education
* BMI between 19 and 30

Exclusion Criteria:

* Diagnosed medical condition
* women who are nursing, pregnant, or plan to become pregnant within 3 months
* History of psychotic disorder or family history of psychotic disorder

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Profile of Mood States (POMS) | End of study (Baseline - time 0 and approximately 8 weeks later)
  The POMS measures individuals' mood states. This is a validated scale to measure positive and negative mood states. The POMS contains 30 items and assesses six identified mood factors: Tension-Anxiety, Depression-Ejection, Anger- Hostility, Vigor-Activity, Fatigue-Inertia, and Confusion-Bewilderment. Scoring of the instrument provides a global score of 0 to 120 or individual domain scores. Lower scores indicate better mood state. The POMS brief form is a simple self-rating instrument.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Matthew Bona, Chicago, Illinois
  - University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bershad AK, Preller KH, Lee R, Keedy S, Wren-Jarvis J, Bremmer MP, de Wit H. Preliminary Report on the Effects of a Low Dose of LSD on Resting-State Amygdala Functional Connectivity. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Apr;5(4):461-467. doi: 10.1016/j.bpsc.2019.12.007. Epub 2019 Dec 20. PMID 32033922
- [Derived] Bershad AK, Schepers ST, Bremmer MP, Lee R, de Wit H. Acute Subjective and Behavioral Effects of Microdoses of Lysergic Acid Diethylamide in Healthy Human Volunteers. Biol Psychiatry. 2019 Nov 15;86(10):792-800. doi: 10.1016/j.biopsych.2019.05.019. Epub 2019 Jun 3. PMID 31331617